CLINICAL TRIAL: NCT01565148
Title: A Randomized, Multi-center, Phase II Study of the Safety, Tolerability, and Bioactivity of Repeated Intravitreal Injections of iCo-007 as Monotherapy or in Combination With Ranibizumab or Laser Photocoagulation in the Treatment of Diabetic Macular Edema With Involvement of the FoveAL Center (the iDEAL Study)
Brief Title: A Randomized, Multi-center, Phase II Study of the Safety, Tolerability and Bioactivity of Repeated Intravitreal Injections of iCo-007 as Monotherapy or in Combination With Ranibizumab or Laser Photocoagulation in the Treatment of Diabetic Macular Edema (the iDEAL Study)
Acronym: iDEAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient's disease progressed and Vision Dropped which led to exit from the study
Sponsor: Johns Hopkins University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); iCo Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010-007-03-DME
Record Dates: First submitted 2012-03-15; First posted 2012-03-28 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema (DME)
MeSH Terms: interventions — Lasers; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Drug: iCo-007 350 mcg
  iCo-007 (350 μg) as an intravitreal injection at baseline followed by another iCo-007 dose (350 μg) at month 4
  Interventions: Drug: iCo-007 350 mcg
- Group 2 (Experimental): Drug: iCo-007 700 mcg
  iCo-007 (700 μg) as an intravitreal injection at baseline followed by another iCo-007 dose (700 μg) at month 4
  Interventions: Drug: iCo-007 700 mcg
- Group 3 (Experimental): Drug: iCo-007 350 mcg and Laser
  iCo-007 (350 μg) as an intravitreal injection at baseline followed 7 days later by laser photocoagulation. At M4, intravitreal injection of iCo-007 (350 μg) will be given as mandatory treatment. If the eye also meets retreatment criteria, it will also receive the second laser photocoagulation
  Interventions: Drug: iCo-007 350 mcg and Laser
- Group 4 (Experimental): Drug: Ranibizumab and iCo-007 350 mcg
  Ranibizumab (0.5 mg) intravitreal injection at baseline followed by iCo-007 (350 μg) intravitreal injection 2 weeks later; re-treatment with ranibizumab (0.5 mg) mandatory at M4 followed by iCo-007 (350 μg) 2 weeks later
  Interventions: Drug: Ranibizumab and iCo-007 350 mcg

INTERVENTIONS:
Drug: iCo-007 350 mcg — iCo-007 (350 μg) as an intravitreal injection at baseline followed by another iCo-007 dose (350 μg) at month 4
  Other Names: Group 1
  Arms: Group 1
Drug: iCo-007 700 mcg — iCo-007 (700 μg) as an intravitreal injection at baseline followed by another iCo-007 dose (700 μg) at month 4
  Other Names: Group 2
  Arms: Group 2
Drug: iCo-007 350 mcg and Laser — iCo-007 (350 μg) as an intravitreal injection at baseline followed 7 days later by laser photocoagulation. At M4, intravitreal injection of iCo-007 (350 μg) will be given as mandatory treatment. If the eye also meets retreatment criteria, it will also receive the second laser photocoagulation
  Other Names: Group 3
  Arms: Group 3
Drug: Ranibizumab and iCo-007 350 mcg — Ranibizumab (0.5 mg) intravitreal injection at baseline followed by iCo-007 (350 μg) intravitreal injection 2 weeks later; re-treatment with ranibizumab (0.5 mg) mandatory at M4 followed by iCo-007 (350 μg) 2 weeks later
  Other Names: Group 4
  Arms: Group 4

SUMMARY:
* To assess the safety of repeated iCo-007 intravitreal injections in treatment of subjects with diabetic macular edema as monotherapy and in combination with ranibizumab or laser photocoagulation
* To assess the change in visual acuity and retinal thickness on optical coherence tomography (OCT) from baseline to month 8 and month 12

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Have diabetes mellitus type I or II (insulin or non-insulin dependent) with HbA1c ≥5.5% and HbA1c ≤13%; have non-proliferative diabetic retinopathy, or inactive proliferative diabetic retinopathy, or proliferative diabetic retinopathy with a reasonable expectation that panretinal photocoagulation will not be required during the study follow-up period
* Have diabetic macular edema with central subfield thickness of ≥250 microns (confirmed by Stratus Time-Domain(TD) OCT
* Have best corrected visual acuity (ETDRS) that is Snellen equivalent of

  * 20/32 and ≥20/320, inclusive
* Be willing and able to sign an approved written informed consent. If a patient has a central nervous system disorder (i.e. dementia) that will not allow him/her to understand the consent independently, the patient will not be allowed to join the study
* Be able to attend all scheduled study visits
* Women who are not lactating or pregnant and are willing to use adequate contraception during the study period, if appropriate

Exclusion Criteria:

* Have macular or perimacular edema secondary to an etiology other than diabetes
* Have concurrent retinal diseases other than diabetic retinopathy
* Have additional ocular diseases compromising visual acuity and/or interfering with study assessments; patients who have glaucoma but deemed stable (intraocular pressure ≤ 25 mmHg at screening) on medications or status post surgery, may participate in the study
* Participant has a history of prior pars plana vitrectomy
* Subjects with significant cataract or or posterior capsular opacification that may need intervention within one year or vitreous opacity that hinder study assessment (i.e.fundus examination) which requires intervention within a year
* Subjects who have DME with severe capillary non-perfusion (avascular zone diameter >1,000 microns)
* Have an allergy to fluorescein dye
* Have terminal renal disease (on active kidney dialysis), cerebral vascular accident(including TIA), myocardial infarction or congestive heart disease within 6 months of study enrollment, liver damage (2x upper limit of normal range for aspartate aminotransferase (AST), Alanine aminotransferase (ALT) or total bilirubin). Patients who may have received renal transplant in the past and now have stable renal function, may participate in the study
* Subjects with systolic blood pressure higher than 180 mm Hg or diastolic above 100 mm Hg, with or without anti-hypertensive treatment
* Have a history of panretinal photocoagulation (PRP) in the study eye within 3 months of study entry or are likely to have PRP in the study eye during study participation
* Had macular photocoagulation or ocular surgery within 3 months of study entry in the study eye
* Received intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 3 months of study entry or anti-angiogenic drugs (pegaptanib sodium, ranibizumab, bevacizumab, VEGF-TRAP, protein kinase C inhibitor, etc.) within 2 months of study entry; history of usage of topical or systemic steroids within 3 months of study entry is not an exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana V. Do, MD, Principal Investigator — Stanley M Truhlsen Eye Institute, University of Nebraska Medical Center; Robert Wong, MD, Principal Investigator — Austin Retina Associates; Michael J. Tolentino, MD, Principal Investigator — Center for Retina Macula Disease; Prema Abraham, MD, Principal Investigator — Black Hills Regional Eye Institute; Eugene Lit, MD, Principal Investigator — East Bay Retina Institute; Michael J. Elman, MD, Principal Investigator — Elman Retina Group; Thomas A. Barnard, MD, Principal Investigator — Florida Retina Institute; Thomas A. Ciulla, MD, Principal Investigator — Midwest Eye Institute; Richard B. Rosen, MD, Principal Investigator — New York Eye and Ear Infirmary; Henry L. Hudson, MD, Principal Investigator — Retina Centers, P.C.; Pravin Dugel, MD, Principal Investigator — Retina Consultants of Arizona; Gregg T. Kokame, MD, Principal Investigator — Retina Consultants of Hawaii, Pali Momi Medical Center; David M. Brown, MD, Principal Investigator — Retina Consultants Houston; Larry S. Halperin, MD, Principal Investigator — Retina Group of Florida; Goergios Papastergio, MD, Principal Investigator — Retina Institute of Hawaii; Ron P. Gallemore, MD. PhD, Principal Investigator — Retina Macula Institute; Brian B. Berger, MD, Principal Investigator — Retina Research Center; Homayoun Tabandeh, MD, Principal Investigator — Retina Vitreous Associates; Dennis M. Marcus, MD, Principal Investigator — Southeast Retina; Robert S. Wirthlin, MD, Principal Investigator — Spokane Eye Clinic; David Callanan, MD, Principal Investigator — Texas Retina Associates in Arlington; Karl G. Csaky, MD, PhD, Principal Investigator — Texas Retina Associates in Dallas; Surendar Purohit, MD, Principal Investigator — TLC Eye Care & Laser Center; Victor H. Gonzalez, MD, Principal Investigator — Valley Retina Institute; Louis Glazer, MD, Principal Investigator — Vitreo-Retinal Associates; Dean Eliott, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary, Harvard Medical School
Locations (1):
- Stanley M Truhlsen Eye Institute, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab and iCo-007 350 mcg: Ranibizumab Plus iCo-007 350 mcg: Ranibizumab (0.5 mg) intravitreal injection at baseline followed by iCo-007 (350 μg) intravitreal injection 2 weeks later; re-treatment with ranibizumab (0.5 mg) mandatory at M4 followed by iCo-007 (350 μg) 2 weeks later
Period: Overall Study
Arm/Group | iCo-007 350 mcg | iCo-007 700 mcg | iCo-007 350 mcg and Laser | Ranibizumab and iCo-007 350 mcg
Started | 47 | 46 | 47 | 45
Completed | 32 | 31 | 40 | 32
Not Completed | 15 | 15 | 7 | 13
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 4 | 4 | 0 | 3
Not completed — Rescue Therapy | 8 | 5 | 5 | 8
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3: iCo-007 350 mcg Plus Laser: iCo-007 (350 μg) as an intravitreal injection at baseline followed 7 days later by laser photocoagulation. At M4, intravitreal injection of iCo-007 (350 μg) will be given as mandatory treatment. If the eye also meets retreatment criteria, it will also receive the second laser photocoagulation
- Group 4: Ranibizumab Plus iCo-007 350 mcg: Ranibizumab (0.5 mg) intravitreal injection at baseline followed by iCo-007 (350 μg) intravitreal injection 2 weeks later; re-treatment with ranibizumab (0.5 mg) mandatory at M4 followed by iCo-007 (350 μg) 2 weeks later
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 47 | 46 | 47 | 45 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.91) | 62.8 (9.7) | 61.4 (9.72) | 61.2 (7.29) | 62.2 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 19 | 20 | 17 | 83
  Male | 20 | 27 | 27 | 28 | 102
Baseline Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: Letters] | 57.9 (12.3) | 58.7 (12.49) | 59.8 (13.78) | 61.5 (14.03) | 59.3 (13.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in VA From Baseline to Month 8
Description: The primary efficacy variable is the change in visual acuity (mean change in number of letters) from baseline to month 8
Time Frame: Baseline to month 8
Population: The results are from the participants which completed the primary end point and for which the data is available.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 28 | 26 | 36 | 29
Letters | -12.07 (18.20) | -24.46 (24.02) | -15.22 (24.62) | -18.28 (30.45)

2. Secondary Outcome: Number of Participants in a Given Study Arm Experiencing the Same Drug-related Serious Adverse Event as a Measure of Safety and Tolerability
Description: Safety of repeated iCo-007 intravitreal injections in treatment of subjects with Diabetic Macular Edema (DME) as monotherapy and in combination with ranibizumab or laser photocoagulation. Serious consideration will be given if 2 or more patients in a particular treatment arm experience the same drug-related serious adverse event;
Time Frame: Baseline to month 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 47 | 46 | 47 | 45
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in VA From Baseline to Month 12
Description: The primary efficacy variable is the change in visual acuity (mean change in number of letters) from baseline to month 12
Time Frame: Baseline to month 12
Population: The study was terminated prior to month 12. No data was collected and 0 participants were analyzed at month 12
Arm/Group | iCo-007 350 mcg | iCo-007 700 mcg | iCo-007 350 mcg and Laser | Ranibizumab and iCo-007 350 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Retinal Thickness Measured by OCT From Baseline to Month 8
Description: Group 1
Time Frame: Baseline to month 8
Population: Some participants opted out of the month 8 OCT.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 25 | 22 | 29 | 22
microns | -70.68 (176.31) | -160.22 (177.36) | -54.17 (125.35) | -92.10 (185.49)

5. Secondary Outcome: Change in Retinal Thickness Measured
Description: measured by OCT
Time Frame: Baseline to month 12
Population: The study was terminated prior to month 12. No data was collected and 0 participants were analyzed at month 12
Arm/Group | iCo-007 350 mcg | iCo-007 700 mcg | iCo-007 350 mcg and Laser | Ranibizumab and iCo-007 350 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Duration of iCo-007 Treatment Effect
Description: treatment effect as measured by VA and OCY thickness
Time Frame: Baseline to month 12
Population: The study was terminated prior to month 12. No data was collected and 0 participants were analyzed at month 12
Arm/Group | iCo-007 350 mcg | iCo-007 700 mcg | iCo-007 350 mcg and Laser | Ranibizumab and iCo-007 350 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Peak Plasma Concentration (Cmax)of iCo-007 After Multiple Injections
Description: cmax
Time Frame: Baseline to month 12
Population: The study was terminated prior to month 12. No data was collected and 0 participants were analyzed at month 12
Arm/Group | iCo-007 350 mcg | iCo-007 700 mcg | iCo-007 350 mcg and Laser | Ranibizumab and iCo-007 350 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 1/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 5/47 | 9/46 | 5/47 | 15/45
Other Adverse Events (participants affected / at risk) | 32/47 | 35/46 | 36/47 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=47) | Group 2 (N=46) | Group 3 (N=47) | Group 4 (N=45)
Ocular Adverse Events (Eye disorders) | 2 (2) | 4 (4) | 3 (3) | 7 (7)
Non-Ocular Adverse Events (General disorders) | 3 (3) | 5 (5) | 2 (2) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=47) | Group 2 (N=46) | Group 3 (N=47) | Group 4 (N=45)
Other Adverse Events - Ocular (Eye disorders) | 28 (107) | 32 (119) | 29 (88) | 34 (99)
Other Adverse Events - Systemic (General disorders) | 20 (58) | 23 (63) | 23 (45) | 22 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No